CLINICAL TRIAL: NCT05954442
Title: An Open, Randomized Phase III Study of Everolimus With Investigator's Choice of Chemotherapy Versus Chemotherapy in The First-Line Treatment of Luminal Androgen Receptor (LAR) Subtype With PI3K/AKT/mTOR Pathway Mutation of Locally Recurrent Inoperable or Metastatic Triple-Negative Breast Cancer (BCTOP-T-M03)
Brief Title: Everolimus With Investigator's Choice of Chemotherapy in Advanced Triple-Negative Breast Cancer (TNBC) With Luminal Androgen Receptor (LAR) Subtype
Acronym: BCTOP-T-M03
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N058
Record Dates: First submitted 2023-07-13; First posted 2023-07-20 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Triple Negative Breast Cancer; Metastatic Breast Cancer; Mutation
Keywords: triple negative breast cancer; metastatic breast cancer; PI3K/AKT/mTOR mutation
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Everolimus plus Investigator's Choice of Chemotherapy
  Interventions: Drug: Everolimus; Drug: Investigator's Choice of Chemotherapy
- Arm B (Active Comparator): Investigator's Choice of Chemotherapy
  Interventions: Drug: Investigator's Choice of Chemotherapy

INTERVENTIONS:
Drug: Everolimus — Everolimus is a kind of mTOR inhibitors which has been approved to use in several kinds of cancers, especially in metastatic breast cancer .
  Other Names: Afinitor
  Arms: Arm A
Drug: Investigator's Choice of Chemotherapy — Investigator's choice of chemotherapy means the chemotherapy chosen by investigators/doctors to treat metastatic triple negative breast cancer, including nab-paclitaxel, capecitabine, eribulin, carboplatin, vinorelbine, or utidelone.
  Other Names: ICC

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of investigator's choice of chemotherapy, either alone or in combination with everolimus, in treating patients with locally recurrent inoperable or metastatic triple-negative breast cancer, luminal androgen receptor (LAR) subtype with PI3K/AKT/mTOR (PAM) pathway mutation, as the first-line treatment.

DETAILED DESCRIPTION:
Eligible participants will be those diagnosed with estrogen receptor (ER)-negative [Immunohistochemistry (IHC) ER positive <1% ) , progesterone receptor (PR) negative(IHC PR positive <1% ) , and human epidermal growth factor receptor 2 (HER2)-negative [IHC 0 or +; or IHC ++, Fluorescence in situ hybridization (FISH) -], LAR subtype with PAM pathway mutation locally recurrent inoperable or metastatic breast cancer, who have received no prior chemotherapy, targeted therapy or other treatments.

The study is aimed to evaluate the efficacy of investigator's choice (ICC) of chemotherapy (nab-paclitaxel, capecitabine, eribulin, carboplatin, vinorelbine, or utidelone) either alone or in combination with everolimus. This study aims to see if everolimus plus chemotherapy allows patients to live longer without the cancer getting worse, or simply to live longer, compared to patients receiving investigator's choice of chemotherapy. This study is also looking to see how the treatment and the cancer affects patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to meet all of the following conditions

  * Patients must be ≥18 and ≤ 70 years of age;
  * Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
  * The expected survival is more than 3 months;
  * Pathologically confirmed breast cancer is triple negative breast cancer (IHC ER < 1%, PR<1%, HER2 0 OR +, if HER2++, FISH negative), and LAR subtype with mutation in PAM pathway;
  * Recurrent or metastatic breast cancer; Patients with local recurrence need to be confirmed by the investigator that radical surgical resection is not possible;.
  * No prior therapy (chemotherapy, targeted therapy, etc.) for advanced or metastatic breast cancer;
  * Patients with at least one lesion (measurable and/or unmeasurable) that has not previously received radiation therapy can be accurately evaluated by CT/MRI at baseline and can be evaluated repeatedly according to RECIST 1.1;
  * The functions of the main organs are basically normal, and the following conditions are met:

    1. Blood routine examination standards should meet: HB≥90g/L (no blood transfusion within 14 days); ANC≥1.5×109/L; PLT≥75×109/L;
    2. Biochemical examination shall meet the following standards: TBIL≤1.5× upper limit of normal value(ULN); alanine aminotransferase (ALT) and AST≤3 x ULN; In case of liver metastasis, ALT and AST≤5×ULN; Serum Cr ≤1×ULN, endogenous creatinine clearance > 50ml/min (Cockcroft-Gault formula);
  * Patients have not received radiotherapy, endocrine therapy, molecular targeted therapy, or surgery within 3 weeks prior to study initiation, and have recovered from acute toxic effects of prior treatment (if surgery is present, the wound has fully healed); No peripheral neuropathy or grade I peripheral neurotoxicity;
  * Fertile female are required to use a medically approved contraceptive during study treatment and for at least 3 months after the last use of the study drug;
  * Patients voluntarily join the study, sign the informed consent, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

* Patients with any of the following conditions were excluded from the study:

  * Patients with known central nervous system metastasis or history of central nervous system metastasis prior to screening. For patients with clinically suspected central nervous system metastasis, enhanced CT or enhanced MRI must be performed within 28 days before the first dose to rule out central nervous system metastasis.
  * A history of clinically significant or uncontrolled heart disease, including congestive heart failure, angina pectoris, myocardial infarction within the last 6 months, or ventricular arrhythmia;
  * Persistent grade ≥1 adverse events due to previous treatment. The exception to this is hair loss or something the researchers believe should not be ruled out. Such cases should be clearly documented in the investigator's notes;
  * Major surgery was performed within 3 weeks of the first course of trial treatment (except for minor outpatient surgery, such as placement of vascular access);
  * Pregnant or lactating patients;
  * Other malignancies within the previous 5 years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma, or skin squamous cell carcinoma;
  * Inability to swallow, chronic diarrhea and intestinal obstruction, there are many factors affecting drug use and absorption;
  * There is a third space effusion that cannot be controlled by drainage or other methods (such as excessive pleural fluid and ascites);
  * Participated in other anti-tumor drug clinical trials within 4 weeks before taking the study drug for the first time;
  * Long-term unhealed wounds or incomplete healing fractures;
  * Patients with known Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection active phase or hepatitis B DNA≥500, or chronic phase with abnormal liver function;
  * Allergic physique, or known allergic history of the drug components of this program; Or allergic to other monoclonal antibodies;
  * The investigator does not consider the patient suitable for participation in any other circumstances of the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Approximately 3 years
  The interval from randomization until the first occurrence of disease progression (according to RECIST 1.1) or death from any cause, which ever occurs first.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Approximately 3 years
  The proportion of participants who have a complete response (CR) or partial response (PR) according to RECIST 1.1.
Duration of response (DoR) | Approximately 3 years
  The interval from date of first detection of objective response until the first occurrence of disease progression (according to RECIST 1.1) or death from any cause, which ever occurs first.
Disease control rate (DCR) | Approximately 3 years
  The proportion of participants with complete response, partial response, and stable disease for more than 4 weeks in which response can be evaluated.
Overall survival (OS) | Approximately 3 years
  The interval from randomization until the date of death due to any cause.
Safety and tolerability | Approximately 3 years
  Number of adverse events according to NCI-CTCAE Version 5.0 per each treatment arm
Number of participants with patient reported outcome (PRO) | Approximately 3 years
  A report directly from a patient about his or her health or life quality by EORTC Core Quality of Life questionnaire (EORTC QLQ-C30). EORTC QLQ-C30 is a 30-item questionnaire and 28 out of 30 items are scored on a 4-point Likert response scale: 1 = not at all, 2 = a little, 3 = quite a bit, and 4 = very much. The EORTC QLQ-C30 scale scores range from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China